CLINICAL TRIAL: NCT03039205
Title: Evaluation of Platelet Aggregation and Adenosine Levels in Patients With Coronary Artery Disease and Chronic Kidney Dysfunction Taking Dual Antiplatelet Therapy With Aspirin and Clopidogrel or Ticagrelor
Brief Title: Platelet Aggregation in Patients With Coronary Artery Disease and Kidney Dysfunction Taking Clopidogrel or Ticagrelor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Jose Carlos Nicolau, Director, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FAPESP 2014/01021-4; 4086/14/066 (Other: CAPPesq)
Record Dates: First submitted 2017-01-23; First posted 2017-02-01 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Platelet Aggregation; Adenosine; Coronary Artery Disease; Kidney Dysfunction; Antiplatelet Therapy
Keywords: Platelet aggregation; Adenosine; Coronary artery disease; Kidney dysfunction; Ticagrelor; Clopidogrel
MeSH Terms: conditions — Coronary Artery Disease | interventions — Clopidogrel; Ticagrelor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Chronic kidney dysfunction Clopidogrel (Active Comparator): Patients with creatinine clearance <60ml/min/m2 (estimated by MDRD formula) randomized to clopidogrel group
  Interventions: Drug: Clopidogrel
- Chronic kidney dysfunction Ticagrelor (Active Comparator): Patients with creatinine clearance <60ml/min/m2 (estimated by MDRD formula) randomized to ticagrelor group
  Interventions: Drug: Ticagrelor
- Normal kidney function Clopidogrel (Active Comparator): Patients with creatinine clearance ≥60ml/min/m2 (estimated by MDRD formula) randomized to clopidogrel group
  Interventions: Drug: Clopidogrel
- Normal kidney function Ticagrelor (Active Comparator): Patients with creatinine clearance ≥60ml/min/m2 (estimated by MDRD formula) randomized to ticagrelor group
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Clopidogrel — Clopidogrel 600 mg loading dose + 75 mg q.d. for 7 to 9 days
  Other Names: Plavix
  Arms: Chronic kidney dysfunction Clopidogrel; Normal kidney function Clopidogrel
Drug: Ticagrelor — Ticagrelor 180 mg loading dose + 90 mg b.i.d. for 7 to 9 days
  Other Names: Brilinta
  Arms: Chronic kidney dysfunction Ticagrelor; Normal kidney function Ticagrelor

SUMMARY:
About 35% of patients hospitalized with Acute Coronary Syndromes (ACS) have some degree of renal dysfunction. Chronic kidney disease (CKD) is not only associated to worse prognosis in ACS patients, but leads also to an increased risk of bleeding, which may importantly influence the risk-benefit ratio of antiplatelet therapy in this population. The responsible mechanisms for increased rate of ischemic events in this population are not completely elucidated.

Antiplatelet therapy is of paramount importance in the treatment of ACS, but its benefit in CKD patients is not well established. This population is often excluded or underrepresented in large clinical trials, and the indication of antiplatelet therapy is often extrapolated from studies in patients with preserved renal function. In recent meta-analysis, Palmer et al. sought to evaluate the benefits and risks of antiplatelet agents in patients with CKD and concluded that in patients with ACS or scheduled for angioplasty already taking aspirin, the addition of clopidogrel or glycoprotein IIb / IIIa inhibitors have little or no impact in reducing the incidence of myocardial infarction, death or need for revascularization.

In the PLATO trial, ticagrelor (a new reversible inhibitor of P2Y12 receptor with faster onset of action and greater platelet inhibition) was compared to clopidogrel in patients with high risk ACS and was associated to a 16% risk reduction on the occurrence of death from vascular causes, myocardial infarction, or stroke. In a pre-specified sub-analysis, data from patients with CKD were compared to those obtained from the population with normal renal function and suggests that the benefit of ticagrelor may be even greater in patients with CKD. Two hypotheses were considered to explain these results:

1. Greater and more consistent platelet inhibition achieved with ticagrelor would be more effective in reducing ischemic events in this population at increased thrombotic risk;
2. Pleiotropic effects of ticagrelor besides inhibition of the P2Y12 receptor. Ticagrelor might be associated with an elevation in serum levels of adenosine. This could improve myocardial perfusion through coronary vasodilation, and this effect would be more pronounced in patients with renal dysfunction.

This project aims to validate (or not) these hypotheses, analyzing platelet aggregation and circulating adenosine levels in patients taking dual antiplatelet therapy with aspirin and clopidogrel or ticagrelor.

DETAILED DESCRIPTION:
Previous publications demonstrated that about 35% to 40% of patients hospitalized with Acute Coronary Syndromes (ACS) have some degree of renal dysfunction. On the other hand, chronic kidney disease (CKD) is not only associated to worse prognosis in ACS patients, but leads also to an increased risk of bleeding, which may importantly influence the risk-benefit ratio of antiplatelet therapy in this population. Even at early stages, CKD increases the risk of myocardial infarction and death among different spectra of ACS, and the risk increase is directly proportional to the degree of renal dysfunction. The responsible mechanisms for the increased rate of ischemic events in this population are not completely elucidated. However, accelerated atherosclerosis, oxidative stress, inflammation and increased platelet aggregation, as well as underutilization of therapies such as antithrombotic agents and invasive procedures, are some of the proposed mechanisms.

Antiplatelet therapy is of paramount importance in the treatment of ACS, but its benefit in CKD patients is not well established. The fact that this population is often excluded or underrepresented in large clinical trials, makes the indication for its use be very often extrapolated from studies in patients with preserved renal function.

In recent meta-analysis, Palmer et al. sought to summarize the benefits and risks of antiplatelet agents in patients with CKD, focusing on the occurrence of cardiovascular events (including mortality) and bleeding. The results led them to conclude that: 1) the evidence for the use of antiplatelet agents in patients with CKD and cardiovascular disease is of low quality, 2) in patients with ACS or scheduled for angioplasty already taking acetylsalicylic acid (ASA), the addition of clopidogrel or glycoprotein IIb / IIIa inhibitors have little or no impact in reducing the incidence of myocardial infarction, death or need for revascularization, and 3) there was a significant 40% increase in the incidence of major bleeding.

In the PLATO trial - "Ticagrelor versus Clopidogrel in Patients with Acute Coronary Syndromes" - ticagrelor, a new reversible inhibitor of the P2Y12 receptor with faster onset of action and greater platelet inhibition power was compared to clopidogrel in over 18,000 patients with high risk ACS. In this publication, patients receiving ticagrelor had a 16% risk reduction on the occurrence of primary composite endpoint (death from vascular causes, myocardial infarction or stroke) without significant increase in the incidence of major bleeding. In a secondary outcome analysis, it was found a significant reduction in mortality from vascular causes and mortality from any cause in patients treated with ticagrelor. Among the high-risk criteria used in the selection of patients for this study, a creatinine clearance <60 ml/min/1.73 m2 was included.

In a following article, considering a pre-specified sub-analysis from the PLATO trial, the results of 3,237 patients who had this high-risk criterion were compared to those obtained for the population with normal renal function. The developed comparisons suggest that the benefit of ticagrelor may be even greater in patients with CKD: when considering the MDRD equation to estimate renal function, the hazard-ratio (HR) for the primary outcome of the study was 0.71 for patients with renal impairment (creatinine clearance <60 ml/min/1.73m2) and 0.90 for those without renal dysfunction (p = 0.03 for interaction). Furthermore, the HRs for mortality were, respectively, 0.79 and 0.91 for patients with and without renal dysfunction (P = 0.02 for interaction). Interestingly, no significant difference between groups relatively to major bleeding was observed, and the incidence of dyspnea was higher in the population without renal dysfunction.

Two hypotheses were considered to explain these results. The first suggests that a greater and more consistent platelet inhibition achieved with ticagrelor would be more effective in reducing ischemic events in this population at increased thrombotic risk. The second hypothesis considers possible pleiotropic effects of ticagrelor besides the reversible inhibition of the P2Y12 receptor. Ticagrelor might be associated with an elevation in serum levels of adenosine through the inhibition of its reuptake by erythrocytes and by increased release of adenosine triphosphate (ATP) from the same erythrocytes, subsequently converted in adenosine by ecto-ATPases. An increase in the concentrations of circulating adenosine could improve myocardial perfusion through coronary vasodilation, and this effect would be more pronounced in patients with renal dysfunction.

Thus, this project aims to validate (or not) these hypotheses, analyzing platelet aggregation and circulating adenosine levels in patients taking dual antiplatelet therapy with aspirin and clopidogrel or ticagrelor.

# Safety: as this protocol was designed for a short-term duration, we do not expect to have many adverse events (AE). An AE is any untoward medical occurrence in a participant that does not necessarily have a causal relationship with the study intervention. An AE can therefore be any unfavorable or unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the use of a medical treatment or procedure regardless of whether it is considered related to the medical treatment or procedure. AEs will be reported as soon as possible.

Serious adverse events (SAE) are defined as any untoward medical occurrence that meets any one of the following criteria:

1. Results in death or is life-threatening at the time of the event;
2. Requires inpatient hospitalization, or prolongs a hospitalization;
3. Results in a persistent or significant disability/incapacity;
4. Is a congenital anomaly/birth defect (in a participants offspring); or
5. Is medically judged to be an important event that jeopardized the subject and, for example, required significant measures to avoid one of the above outcomes.

SAEs will be reported within 24 hours of its information received. The causality of SAEs (their relationship to all study treatment/procedures) will be assessed by the investigator(s) and the investigator is responsible for informing the local authorities and ethical committees, of any serious adverse events as per local requirements.

ELIGIBILITY:
Inclusion Criteria:

* Patients in use of aspirin for at least 7 days prior to randomization;
* Documented obstructive coronary artery disease by angiography;
* At least 12 months from the last episode of myocardial infarction (MI);
* Agree to sign the Informed Consent.

Exclusion Criteria:

* Prior ischemic or hemorrhagic stroke;
* Prior intracranial bleeding;
* Use of oral anticoagulant in the past month;
* Use of dual antiplatelet therapy in the last 30 days;
* Use of NSAIDs and / or dipyridamole in the past month;
* Mandatory use of proton pump inhibitor;
* Known platelet dysfunction or platelets <100,000 or >450,000/μL;
* End-stage renal disease undergoing hemodialysis;
* Terminal illness;
* Known liver disease or coagulation disorder;
* Known pregnancy, breast-feeding, or intend to become pregnant during the study period;
* Hypersensitivity to clopidogrel, ticagrelor or any excipients;
* Refusal to sign the Informed Consent;
* Active pathological bleeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2019-12-19 (Actual)

PRIMARY OUTCOMES:
Platelet aggregation evaluated by VerifyNow® P2Y12 (difference between clopidogrel and ticagrelor) in patients with and without renal dysfunction randomized to treatment with either clopidogrel or ticagrelor | 8 days (±1)
  Compare the level of inhibition of platelet aggregation evaluated by VerifyNow® P2Y12 (difference between clopidogrel and ticagrelor) in patients with coronary artery disease with and without renal dysfunction undergoing treatment with ASA in combination with clopidogrel or ticagrelor.

SECONDARY OUTCOMES:
Adenosine plasma concentration evaluated by isocratic high-performance liquid chromatographic technique, in patients with and without renal dysfunction randomized to treatment with either clopidogrel or ticagrelor. | 8 days (±1)
  Compare adenosine plasma concentration evaluated by isocratic high-performance liquid chromatographic technique, in patients with coronary artery disease with and without renal dysfunction undergoing treatment with ASA in combination with clopidogrel or ticagrelor.
Platelet aggregation (difference between clopidogrel and ticagrelor) evaluated by Multiple electrode platelet aggregometry (Multiplate®) in patients with and without renal dysfunction randomized to treatment with either clopidogrel or ticagrelor | 8 days (±1)

OTHER OUTCOMES:
Lipoprotein-a - Lp(a) concentration in the groups with or without renal dysfunction | 8 days (±1)
Hemoglobin concentration in the groups with or without renal dysfunction | 8 days (±1)
Leukocytes concentration in the groups with or without renal dysfunction | 8 days (±1)
Platelet count in the groups with or without renal dysfunction | 8 days (±1)
Prothrombin time in the groups with or without renal dysfunction | 8 days (±1)
Activated partial thromboplastin time in the groups with or without renal dysfunction | 8 days (±1)
Creatinine concentration in the groups with or without renal dysfunction | 8 days (±1)
Urea concentration in the groups with or without renal dysfunction | 8 days (±1)
Total and free cholesterol concentration in the groups with or without renal dysfunction | 8 days (±1)
Free fatty acids concentration in the groups with or without renal dysfunction | 8 days (±1)
Cholesterol-ester transfer protein activity in the groups with or without renal dysfunction | 8 days (±1)
LDL-cholesterol concentration in the groups with or without renal dysfunction | 8 days (±1)
HDL cholesterol concentration, size and transport in the groups with or without renal dysfunction | 8 days (±1)
Triglycerides concentration in the groups with or without renal dysfunction | 8 days (±1)
Fasting glucose concentration in the groups with or without renal dysfunction | 8 days (±1)
Glycated hemoglobin in the groups with or without renal dysfunction | 8 days (±1)
Ultra-sensitive C-reactive protein (usCRP) concentration in the groups with or without renal dysfunction | 8 days (±1)
Interleukin-6 (IL-6) concentration in the groups with or without renal dysfunction | 8 days (±1)
Plasminogen activator inhibitor (PAI-1) concentration in the groups with or without renal dysfunction | 8 days (±1)
Compare platelet aggregation (VerifyNow and Multiplate) and adenosine plasma concentration in the following subgroups: gender (male x female) | 8 days (±1)
Compare platelet aggregation (VerifyNow and Multiplate) and adenosine plasma concentration in the following subgroups: diabetes (present or absent) | 8 days (±1)
Compare platelet aggregation (VerifyNow and Multiplate) and adenosine plasma concentration in the following subgroups: smoking status (yes or no) | 8 days (±1)
Compare platelet aggregation (VerifyNow and Multiplate) and adenosine plasma concentration in the following subgroups: hypertension (presence or absence) | 8 days (±1)
Compare platelet aggregation (VerifyNow and Multiplate) and adenosine plasma concentration in the following subgroups: levels of LDL (<70 or ≥ 70 mg / dl) | 8 days (±1)
Compare platelet aggregation (VerifyNow and Multiplate) and adenosine plasma concentration in the following subgroups: elderly and non-elderly (≥ or <75 years) | 8 days (±1)
Compare platelet aggregation (VerifyNow and Multiplate) and adenosine plasma concentration in the following subgroups: weight (<or ≥ 60 kg) | 8 days (±1)
Compare platelet aggregation (VerifyNow and Multiplate) and adenosine plasma concentration in the following subgroups: body mass index (<30 or ≥ 30kg/m2) | 8 days (±1)
Compare platelet aggregation (VerifyNow and Multiplate) and adenosine plasma concentration in the following subgroups: creatinine clearance (≥60 ml/min, <60 to 30 ml/min and <30 ml/min). | 8 days (±1)
Analyze the influence of angiotensin converting enzyme inhibitors or angiotensin receptor subtype 1 (AT1) blockers on platelet aggregation (VerifyNow and Multiplate) and adenosine plasma concentration | 8 days (±1)
Analyze the influence of oral hypoglycemic agents on platelet aggregation (VerifyNow and Multiplate) and adenosine plasma concentration | 8 days (±1)
Analyze the influence of insulin on platelet aggregation (VerifyNow and Multiplate) and adenosine plasma concentration | 8 days (±1)
Analyze the influence of beta-blockers on platelet aggregation (VerifyNow and Multiplate) and adenosine plasma concentration | 8 days (±1)
Analyze the influence of proton pump inhibitors (PPI) on platelet aggregation (VerifyNow and Multiplate) and adenosine plasma concentration | 8 days (±1)
Analyze, in the studied groups with or without renal dysfunction, the incidence of dyspnea. | 8 days (±1)

CONTACTS AND LOCATIONS:
Overall Officials: José C Nicolau, M.D. / PhD, Study Chair — Heart Institute (InCor) / University of São Paulo; André Franci, M.D., Principal Investigator — Heart Institute (InCor) / University of São Paulo
Locations (1):
- Instituto do Coração (InCor) - Hospital das Clínicas da FMUSP, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Al Suwaidi J, Reddan DN, Williams K, Pieper KS, Harrington RA, Califf RM, Granger CB, Ohman EM, Holmes DR Jr; GUSTO-IIb, GUSTO-III, PURSUIT. Global Use of Strategies to Open Occluded Coronary Arteries. Platelet Glycoprotein IIb/IIIa in Unstable Angina: Receptor Suppression Using Integrilin Therapy; PARAGON-A Investigators. Platelet IIb/IIIa Antagonism for the Reduction of Acute coronary syndrome events in a Global Organization Network. Prognostic implications of abnormalities in renal function in patients with acute coronary syndromes. Circulation. 2002 Aug 20;106(8):974-80. doi: 10.1161/01.cir.0000027560.41358.b3. PMID 12186803
- [Background] Freeman RV, Mehta RH, Al Badr W, Cooper JV, Kline-Rogers E, Eagle KA. Influence of concurrent renal dysfunction on outcomes of patients with acute coronary syndromes and implications of the use of glycoprotein IIb/IIIa inhibitors. J Am Coll Cardiol. 2003 Mar 5;41(5):718-24. doi: 10.1016/s0735-1097(02)02956-x. PMID 12628712
- [Background] Anavekar NS, McMurray JJ, Velazquez EJ, Solomon SD, Kober L, Rouleau JL, White HD, Nordlander R, Maggioni A, Dickstein K, Zelenkofske S, Leimberger JD, Califf RM, Pfeffer MA. Relation between renal dysfunction and cardiovascular outcomes after myocardial infarction. N Engl J Med. 2004 Sep 23;351(13):1285-95. doi: 10.1056/NEJMoa041365. PMID 15385655
- [Background] Best PJ, Lennon R, Ting HH, Bell MR, Rihal CS, Holmes DR, Berger PB. The impact of renal insufficiency on clinical outcomes in patients undergoing percutaneous coronary interventions. J Am Coll Cardiol. 2002 Apr 3;39(7):1113-9. doi: 10.1016/s0735-1097(02)01745-x. PMID 11923033
- [Background] Fox CS, Muntner P, Chen AY, Alexander KP, Roe MT, Cannon CP, Saucedo JF, Kontos MC, Wiviott SD; Acute Coronary Treatment and Intervention Outcomes Network registry. Use of evidence-based therapies in short-term outcomes of ST-segment elevation myocardial infarction and non-ST-segment elevation myocardial infarction in patients with chronic kidney disease: a report from the National Cardiovascular Data Acute Coronary Treatment and Intervention Outcomes Network registry. Circulation. 2010 Jan 26;121(3):357-65. doi: 10.1161/CIRCULATIONAHA.109.865352. Epub 2010 Jan 11. PMID 20065168
- [Background] Ezekowitz J, McAlister FA, Humphries KH, Norris CM, Tonelli M, Ghali WA, Knudtson ML; APPROACH Investigators. The association among renal insufficiency, pharmacotherapy, and outcomes in 6,427 patients with heart failure and coronary artery disease. J Am Coll Cardiol. 2004 Oct 19;44(8):1587-92. doi: 10.1016/j.jacc.2004.06.072. PMID 15489090
- [Background] Antithrombotic Trialists' Collaboration. Collaborative meta-analysis of randomised trials of antiplatelet therapy for prevention of death, myocardial infarction, and stroke in high risk patients. BMJ. 2002 Jan 12;324(7329):71-86. doi: 10.1136/bmj.324.7329.71. PMID 11786451
- [Background] Basra SS, Tsai P, Lakkis NM. Safety and efficacy of antiplatelet and antithrombotic therapy in acute coronary syndrome patients with chronic kidney disease. J Am Coll Cardiol. 2011 Nov 22;58(22):2263-9. doi: 10.1016/j.jacc.2011.08.051. PMID 22093501
- [Background] Palmer SC, Di Micco L, Razavian M, Craig JC, Perkovic V, Pellegrini F, Copetti M, Graziano G, Tognoni G, Jardine M, Webster A, Nicolucci A, Zoungas S, Strippoli GF. Effects of antiplatelet therapy on mortality and cardiovascular and bleeding outcomes in persons with chronic kidney disease: a systematic review and meta-analysis. Ann Intern Med. 2012 Mar 20;156(6):445-59. doi: 10.7326/0003-4819-156-6-201203200-00007. PMID 22431677
- [Background] Wallentin L, Becker RC, Budaj A, Cannon CP, Emanuelsson H, Held C, Horrow J, Husted S, James S, Katus H, Mahaffey KW, Scirica BM, Skene A, Steg PG, Storey RF, Harrington RA; PLATO Investigators; Freij A, Thorsen M. Ticagrelor versus clopidogrel in patients with acute coronary syndromes. N Engl J Med. 2009 Sep 10;361(11):1045-57. doi: 10.1056/NEJMoa0904327. Epub 2009 Aug 30. PMID 19717846
- [Background] James S, Budaj A, Aylward P, Buck KK, Cannon CP, Cornel JH, Harrington RA, Horrow J, Katus H, Keltai M, Lewis BS, Parikh K, Storey RF, Szummer K, Wojdyla D, Wallentin L. Ticagrelor versus clopidogrel in acute coronary syndromes in relation to renal function: results from the Platelet Inhibition and Patient Outcomes (PLATO) trial. Circulation. 2010 Sep 14;122(11):1056-67. doi: 10.1161/CIRCULATIONAHA.109.933796. Epub 2010 Aug 30. PMID 20805430
- [Background] Levey AS, Bosch JP, Lewis JB, Greene T, Rogers N, Roth D. A more accurate method to estimate glomerular filtration rate from serum creatinine: a new prediction equation. Modification of Diet in Renal Disease Study Group. Ann Intern Med. 1999 Mar 16;130(6):461-70. doi: 10.7326/0003-4819-130-6-199903160-00002. PMID 10075613
- [Background] Ohman J, Kudira R, Albinsson S, Olde B, Erlinge D. Ticagrelor induces adenosine triphosphate release from human red blood cells. Biochem Biophys Res Commun. 2012 Feb 24;418(4):754-8. doi: 10.1016/j.bbrc.2012.01.093. Epub 2012 Jan 27. PMID 22306816
- [Background] Montalescot G, Silvain J. Ticagrelor in the renal dysfunction subgroup: subjugated or substantiated? Circulation. 2010 Sep 14;122(11):1049-52. doi: 10.1161/CIRCULATIONAHA.110.974683. Epub 2010 Aug 30. No abstract available. PMID 20805425
- [Background] Park SH, Kim W, Park CS, Kang WY, Hwang SH, Kim W. A comparison of clopidogrel responsiveness in patients with versus without chronic renal failure. Am J Cardiol. 2009 Nov 1;104(9):1292-5. doi: 10.1016/j.amjcard.2009.06.049. PMID 19840579
- [Background] Butler K, Teng R. Pharmacokinetics, pharmacodynamics, and safety of ticagrelor in volunteers with severe renal impairment. J Clin Pharmacol. 2012 Sep;52(9):1388-98. doi: 10.1177/0091270011415526. Epub 2011 Sep 29. PMID 21960668
- [Background] Gurbel PA, Bliden KP, Butler K, Tantry US, Gesheff T, Wei C, Teng R, Antonino MJ, Patil SB, Karunakaran A, Kereiakes DJ, Parris C, Purdy D, Wilson V, Ledley GS, Storey RF. Randomized double-blind assessment of the ONSET and OFFSET of the antiplatelet effects of ticagrelor versus clopidogrel in patients with stable coronary artery disease: the ONSET/OFFSET study. Circulation. 2009 Dec 22;120(25):2577-85. doi: 10.1161/CIRCULATIONAHA.109.912550. Epub 2009 Nov 18. PMID 19923168
- [Background] Storey RF, Angiolillo DJ, Patil SB, Desai B, Ecob R, Husted S, Emanuelsson H, Cannon CP, Becker RC, Wallentin L. Inhibitory effects of ticagrelor compared with clopidogrel on platelet function in patients with acute coronary syndromes: the PLATO (PLATelet inhibition and patient Outcomes) PLATELET substudy. J Am Coll Cardiol. 2010 Oct 26;56(18):1456-62. doi: 10.1016/j.jacc.2010.03.100. PMID 20832963
- [Background] Sibbing D, Braun S, Jawansky S, Vogt W, Mehilli J, Schomig A, Kastrati A, von Beckerath N. Assessment of ADP-induced platelet aggregation with light transmission aggregometry and multiple electrode platelet aggregometry before and after clopidogrel treatment. Thromb Haemost. 2008 Jan;99(1):121-6. doi: 10.1160/TH07-07-0478. PMID 18217143
- [Derived] Natale P, Palmer SC, Saglimbene VM, Ruospo M, Razavian M, Craig JC, Jardine MJ, Webster AC, Strippoli GF. Antiplatelet agents for chronic kidney disease. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD008834. doi: 10.1002/14651858.CD008834.pub4. PMID 35224730
- See also: Isocratic high-performance liquid chromatographic determination of plasma adenosine — http://link.springer.com/article/10.1007/BF02290317